CLINICAL TRIAL: NCT02993146
Title: Phase 1 and Pharmacology Study of Oral 5-Iodo-2-Pyrimidinone-2-Deoxyribose (IPdR) as a Prodrug for IUdR-Mediated Tumor Radiosensitization in Brain Metastases
Brief Title: Ropidoxuridine and Whole Brain Radiation Therapy in Treating Patients With Brain Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01909; NCI-2016-01909 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HP-00067789; 9979 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 9979 (Other: CTEP); UM1CA186686 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2016-12-15 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Hematologic Neoplasms; Brain Neoplasms | interventions — ropidoxuridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ropidoxuridine, WBRT) (Experimental): Patients receive ropidoxuridine PO QD on days 1-28 and undergo WBRT daily for not more than 5 days per week beginning on day 8 for a total of 15 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Drug: Ropidoxuridine; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Ropidoxuridine — Given PO
  Other Names: 5-Iodo-2-pyrimidinone 2' deoxyribonucleoside; 5-Iodo-2-pyrimidinone-2'-deoxyribose; IPdR
Radiation: Whole-Brain Radiotherapy — Undergo WBRT
  Other Names: WBRT; whole-brain radiation therapy

SUMMARY:
This phase I trial studies the side effects and best dose of ropidoxuridine when given together with whole brain radiation therapy in treating patients with cancer that has spread to the brain (brain metastases). Ropidoxuridine may help whole brain radiation therapy work better by making cancer cells more sensitive to the radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a phase 1 dose escalation trial in patients with brain metastases to determine the recommended phase -2 dose of ropidoxuridine (5-iodo-2-pyrimidinone-2'-deoxyribose [IPdR]) when administered alone orally once daily for 7 consecutive days and then concurrently with conventionally fractionated whole brain radiation therapy (WBRT) for additional 21 days.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity to IPdR-mediated radiosensitization.

II. To estimate 6 month intracranial progression-free survival (PFS) in brain metastasis cancer patients who receive daily oral IPdR x 28 days and WBRT.

III. To establish the pharmacokinetics of daily oral dosing of IPdR times 8 days.

IV. To evaluate safety and tolerability of oral IPdR x 28 days and WBRT.

V. To estimate the incidence of delayed neurological toxicity at 2, 4, and 6 months (+/-1 week) post-completion of WBRT (for patients without intracranial progression) including:

Va. Delayed-recall through Hopkins Verbal Learning Test Revised (HVLT-R). Vb. Quality of life as measured by the Functional Assessment of Cancer Therapy-Brain (FACT-BR).

CORRELATIVE OBJECTIVES:

I. To assess for biochemical evidence of IPdR effect in normal tissues (circulating granulocytes) by measuring %IUdR-deoxyribonucleic acid (DNA) cellular incorporation by flow cytometry and high-pressure liquid chromatography (HPLC) analyses as an exploratory biomarker for the following:

Ia. %IUdR-DNA tumor cell incorporation from day 8 extracranial tumor biopsies in brain metastasis cancer patients receiving RP2D doses of IPdR as an exploratory biomarker of tumor radiosensitization using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

Ib. %IUdR-DNA cellular incorporation in patients' circulating granulocytes taken weekly during the 28-day IPdR RP2D dose, on day 29, and week 8 as an exploratory biomarker of IPdR systemic toxicities to bone marrow as measured by serial complete blood count (CBC)/differential values.

OUTLINE: This is a dose escalation study of ropidoxuridine.

Patients receive ropidoxuridine orally (PO) once daily (QD) on days 1-28 and undergo WBRT daily for not more than 5 days per week beginning on day 8 for a total of 15 fractions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 6 months, every 3-4 months for 6 months, and every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy with brain metastases and are being recommended palliative WBRT
* Life expectancy of greater than 2 months to allow completion of study treatment and assessment of dose-limiting toxicity
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Calculated creatinine clearance >= 45 mL/min/1.73 m^2
* Total bilirubin:

  * If no known liver metastases: total bilirubin < 1.5 x institutional upper limit of normal (ULN)
  * If known liver metastases, then: total bilirubin < 2.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]):

  * If no known liver metastases: AST/SGOT and ALT/SGPT both < 2 x ULN
  * If known liver metastases, then: AST/SGOT and ALT/SGPT both < 5 x ULN
* Human immunodeficiency virus (HIV) positive (+) patients with CD4 counts >= 250 cells/mm^3 on anti-viral therapy are eligible for the study
* Negative urine or serum pregnancy test result for females of child bearing potential only; Note: The effects of IPdR on the developing human fetus are unknown; for this reason and because radiation therapy is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of IPdR administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Presence of diffuse lepto or pachy meningeal carcinomatosis (focal/localized involvement from limited meningeal based metastases acceptable), greater than 1 cm mid-line shift, uncal herniation, or severe hemorrhage/hydrocephalous (small intra-lesional hemorrhage or anticipated surgical cavity is acceptable); patients with seizure at presentation who have been started on levetiracetam and have been stable for 48 hours prior to study registration are eligible at the discretion of treating physician
* Patients who have received systemic cytotoxic chemotherapy or approved oral targeted therapy or immunotherapy for 2 weeks, or other investigational agents for 3 weeks (4 half-lives for any oral targeted agents), or radiotherapy to a non-brain site for 2 weeks before initiation of IPdR therapy; patients who have recovered from serious (Common Terminology Criteria for Adverse Events [CTCAE] grade 3 or more higher) to grade 1 or less adverse events from the previous therapies are eligible; prior/current/future hormonal therapy and/or bisphosphonates are permitted with no minimum interval to initiation of study therapy; if indicated, patients can receive palliative radiation therapy to a non-brain site concurrent or immediately post-study treatment with no minimum interval to initiation of study therapy
* Patients must not have received prior whole brain radiation therapy; previous SRS/SRT done at least 3 weeks from the planned start of IPdR therapy is acceptable; SRS/SRT/fractionated boosts or neurosurgery can be performed once the dose limiting toxicity (DLT) assessment has been completed, if felt clinically necessary
* Patients with primary tumors including germ cell tumor, or lymphoma/leukemia
* Patients who are receiving any other investigational agent
* Patients needing more than 8 mg dexamethasone per day at the time of start of WBRT will not be eligible to participate in the study; however, patients will be allowed entry into the study if it is medically safe to reduce the daily dose of dexamethasone to 8 mg or less from the day of the start of WBRT; the dexamethasone dose for such patients may be increased beyond 8 mg per day during the course of treatment if medically necessary; this increased need for dose should be communicated to the study's principal investigator, Dr Mohindra at the University of Maryland
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IPdR
* Uncontrolled intercurrent illness if it would increase the risk of toxicity or limit compliance with study requirements; this includes, but is not limited to, ongoing uncontrolled serious infection requiring intravenous (i.v.) antibiotics, progressive congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because IPdR is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IPdR, breastfeeding should be discontinued if the mother is treated with IPdR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2026-10-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pranshu Mohindra, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (14):
- United States (14):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1A: Patients receive ropidoxuridine 150 mg by mouth on days 1-28 and undergo whole-brain radiotherapy (WBRT) daily, except weekends, for not more than 5 days per week beginning on day 8 for a total of 15 fractions.
- Dose Level 1B: Patients receive ropidoxuridine 300 mg by mouth on days 1-28 and undergo whole-brain radiotherapy (WBRT) daily, except weekends, for not more than 5 days per week beginning on day 8 for a total of 15 fractions.
- Dose Level 2A: Patients receive ropidoxuridine 1200 mg by mouth on days 1-28 and undergo whole-brain radiotherapy (WBRT) daily, except weekends, for not more than 5 days per week beginning on day 8 for a total of 15 fractions.
- Dose Level 2B: Patients receive ropidoxuridine 1800 mg by mouth on days 1-28 and undergo whole-brain radiotherapy (WBRT) daily, except weekends, for not more than 5 days per week beginning on day 8 for a total of 15 fractions.
Period: Overall Study
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Started | 1 | 1 | 7 | 2
Completed | 1 | 1 | 6 | 1
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B | Total
Number analyzed (Participants) | 1 | 1 | 7 | 2 | 11
Age, Continuous [Median (Full Range); unit: years] | 48 [48 to 48] | 50 [50 to 50] | 60 [55 to 73] | 58 [47 to 68] | 58 [47 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 2 | 7
  Male | 1 | 0 | 3 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 7 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 2
  White | 0 | 0 | 7 | 2 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 7 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose Limiting Toxicity
Description: Dose limiting toxicities are protocol-defined, treatment-related adverse events.
Time Frame: Up to week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Number analyzed (Participants) | 1 | 1 | 6 | 1
Participants
  Experienced a dose limiting toxicity | 0 | 0 | 0 | 1
  Did not experience a dose limiting toxicity | 1 | 1 | 6 | 0

2. Secondary Outcome: Number of Participants With Complete Response, Partial Response, Stable Disease or Progressive Disease.
Description: To observe and record anti-tumor activity as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Complete response is no remaining tumor. Partial response is a 30% or greater decrease in overall tumor burden. Progressive disease is a 20% or greater increase in tumor burden. Stable disease is between 20% increase and 30% decrease.
Time Frame: Up to 2 years
Population: Only participants in Part 2 are included in this objective. Data was not collected for participants in Part 1 (DL 1A and 1B).
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Number analyzed (Participants) | 0 | 0 | 6 | 1
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 0 | 0 | 2 | 1
  Progressive Disease | 0 | 0 | 1 | 0
  Not assessed/Unknown | 0 | 0 | 3 | 0

3. Secondary Outcome: Intracranial Disease Status
Description: Intracranial disease status assessed at month 6.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Number analyzed (Participants) | 1 | 1 | 6 | 1
Participants
  Intracranial disease free | 0 | 1 | 1 | 0
  Intracranial disease progression | 1 | 0 | 1 | 1
  Unknown | 0 | 0 | 4 | 0

4. Secondary Outcome: Pharmacokinetics of Oral IPdR
Description: To establish the pharmacokinetics of daily oral dosing of IPdR for 8 days.
Time Frame: At Day 8
Population: Collection not performed.
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Experience Grade 3, 4, or 5 Adverse Events
Description: To establish safety and tolerability of oral IPdR for 28 days with whole brain radiation treatment.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Number analyzed (Participants) | 1 | 1 | 6 | 1
Participants
  Grade 5 adverse events | 0 | 0 | 0 | 0
  Grade 4 adverse events | 0 | 0 | 0 | 0
  Grade 3 adverse events | 0 | 0 | 2 | 1
  Grade 1-2 adverse events | 1 | 1 | 4 | 0

6. Secondary Outcome: Number of Participants With Delayed Neurological Toxicity
Description: To estimate the incidence of delayed neurological toxicity at 2, 4, and 6 months after whole blood radiation treatment.
Time Frame: At 6 months
Population: Assessment not collected
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Dose Level 1A | Dose Level 1B | Dose Level 2A | Dose Level 2B
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1 | 3/7 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 2/7 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 6/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1A (N=1) | Dose Level 1B (N=1) | Dose Level 2A (N=7) | Dose Level 2B (N=1)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1A (N=1) | Dose Level 1B (N=1) | Dose Level 2A (N=7) | Dose Level 2B (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Angioedema R lower lip (Vascular disorders) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0
Aphthous Ulcer (General disorders) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0
Dry dark skin at frontal lobe (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 6 | 0
Fever (General disorders) | 0 | 0 | 0 | 1
Floaters (Eye disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 5 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Increased LDH (Investigations) | 1 | 0 | 0 | 0
Left Knee edema (General disorders) | 1 | 0 | 0 | 0
Leukopenia (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 5 | 0
Numbs gum/less sensation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Scratching (Eye disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrush (Infections and infestations) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Watering eyes (Eye disorders) | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT02993146/Prot_SAP_000.pdf